CLINICAL TRIAL: NCT06776666
Title: Comparison of Pulse Pressure Variation and Central Venous Pressure for Fluid Management Guidance in Intracranial Tumor Surgery
Brief Title: Pulse Pressure Variation Vs. Central Venous Pressure for Fluid Management in Intracranial Tumor Surgery
Acronym: PPV-CVP-FLUID
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Gizem Demirci, Principal investigator, Pamukkale University
Other Study IDs: E-60116787-020-512899; ET-GD-CVP-PPV-FLD-001 (Other: Pamukkale-uni-gd)
Record Dates: First submitted 2024-12-31; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Brain Tumor Adult; Pulse Pressure Variation; Central Venous Pressure; Fluid Management; Brain Surgery
Keywords: Central venous pressure; Fluid management; Brain tumors; Pulse pressure variation; Surgery
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PPV: Patients with intraoperative fluid management according to PPV parameters
- CVP: patients with intraoperative fluid management according to CVP parameters

SUMMARY:
This study investigates the efficacy of pulse pressure variation (PPV) compared to central venous pressure (CVP) in guiding fluid management during intracranial tumor surgeries. Perioperative fluid therapy is critical to prevent complications arising from both hypovolemia (e.g., hypotension, tissue hypoperfusion, ischemia) and hypervolemia (e.g., pulmonary edema, delayed wound healing, infection). Traditional fluid therapy relies on static parameters such as CVP, which have limited sensitivity and specificity. Emerging technologies and dynamic parameters, including PPV and stroke volume variation (SVV), offer higher accuracy in evaluating fluid responsiveness.

This randomized study includes 42 patients, aged 18-65 years, undergoing elective intracranial tumor surgery under general anesthesia. Patients are classified as ASA I-III and are randomized into two groups:

1. Group N: Fluid therapy guided by PPV.
2. Group S: Fluid therapy guided by CVP. The study follows standard perioperative protocols, with PPV (>13%) and CVP (0-6 mmHg) used as primary parameters for fluid administration. Key outcomes include intraoperative fluid requirements (primary) and secondary parameters such as serum lactate levels, incidence of hypotension, brain relaxation scores, and ICU length of stay.

PPV has been shown to be more reliable than CVP in predicting fluid responsiveness, particularly in mechanically ventilated patients with tidal volumes ≥8 mL/kg. However, its efficacy in neurosurgical patients remains underexplored. This study aims to determine if PPV can replace CVP as a superior guide for fluid therapy, enhancing patient outcomes and minimizing complications.

DETAILED DESCRIPTION:
To prevent fluid losses secondary to surgery, fluid therapy should be administered to patients during the preoperative, intraoperative, and postoperative periods. The goal of perioperative fluid therapy is to maintain adequate circulating volume and pressure, avoid dehydration and the adverse effects of excessive fluid administration, and optimize oxygen delivery to tissues to ensure sufficient perfusion. Inadequate fluid administration can result in hypovolemia, leading to complications such as hypotension, tissue hypoperfusion, ischemia, arrhythmias, and renal damage. Conversely, excessive fluid administration can cause hypervolemia-related issues, including fluid accumulation in tissues (especially in the lungs), impaired tissue perfusion, prolonged mechanical ventilation, anastomotic leaks, delayed wound healing, and infections. Postoperative complications can also increase morbidity, mortality, and healthcare costs. Therefore, achieving normovolemia in patients during the perioperative period is of paramount importance.

In traditional fluid therapy, hourly fluid requirements for maintenance and fasting-related deficits are calculated using the '4-2-1' rule (4 mL/kg/hour for the first 10 kg, 2 mL/kg/hour for the next 10 kg, and 1 mL/kg/hour for each kilogram thereafter). Estimated fluid losses from surgical bleeding and evaporation are added to these calculations for replacement. In traditional fluid therapy, intravascular volume is estimated using parameters such as arterial blood pressure, heart rate (HR), and urine output. However, these parameters are influenced by many factors and do not always accurately reflect intravascular volume. Managing patients using these parameters, especially in high-risk surgeries, can result in complications related to hypovolemia and hypervolemia. The lack of an optimal perioperative fluid therapy approach in high-risk surgeries has led to new explorations, including personalized, goal-directed fluid therapy facilitated by advanced technological devices. Studies have shown that personalized, goal-directed fluid therapy improves postoperative outcomes.

Various static parameters have been used to guide fluid therapy to date, one of which is CVP (central venous pressure), commonly employed in clinical practice. The normal range of CVP in the supine position is 0-6 mmHg. A CVP below this range indicates hypovolemia, while a CVP above it suggests hypervolemia. Recent studies have shown that CVP's sensitivity and specificity in detecting fluid deficits are insufficient.

In recent years, dynamic parameters with high sensitivity and specificity, such as PPV (pulse pressure variation) and SVV (stroke volume variation), have been increasingly utilized to assess fluid deficits. Changes in arterial pressure waveforms during respiration are used to evaluate the response to fluid administration. These changes occur during controlled mechanical ventilation. Positive pressure ventilation increases intrathoracic pressure during inspiration, reducing venous return, right ventricular filling volume, and left ventricular stroke volume. During expiration, the effects are reversed. If arterial vasomotor tone and cardiac function remain constant, these changes in stroke volume during positive pressure ventilation are reflected in pulse pressure and systolic blood pressure. In fluid-nonresponsive patients, variations in these dynamic parameters are less than 10%.

In mechanically ventilated, hemodynamically stable, and intubated patients with a tidal volume ≥8 mL/kg, a stroke volume variation (SVV) >10% and a pulse pressure variation (PPV) >13% indicate a fluid deficit.

PPV has been demonstrated to be more reliable than CVP in predicting fluid responsiveness in various studies. However, there are limited studies evaluating the efficacy of PPV in neurosurgical patient populations. Due to the scarcity of studies in the literature, this study aims to compare the efficacy of fluid management guided by PPV and CVP in patients undergoing intracranial tumor surgery. This study aims to evaluate whether PPV can effectively guide fluid therapy and replace CVP in neurosurgical patients undergoing intracranial tumor surgery.

A total of 42 patients aged 18-65 years, undergoing elective intracranial mass surgery under general anesthesia, with an ASA (American Society of Anesthesiologists) physical status classification score of I-III, will be included in the study. Patients with renal failure, mental retardation, arrhythmia, severe cardiopulmonary disease, hemodynamic instability, body mass index (BMI) >40 kg/m², respiratory system compliance (Crs) <30 mL/cmH₂O, use of lactate-producing medications such as metformin, preoperative elevated lactate levels, tumors causing diabetes insipidus, or those refusing the procedure will be excluded from the study. Patients experiencing massive intraoperative bleeding, failing central venous catheter (CVC) placement, or requiring postoperative ventilator support will also be excluded. All procedures to be performed on the study participants will be explained in detail, and informed consent forms will be signed. The invasive procedures, drug applications, and monitoring methods in this study are within the scope of routine practice.

The 42 patients included in the study will be randomized using a computer-generated sampling method into two groups: Group N (n=21), receiving intraoperative fluid management based on PPV (pulse pressure variation) parameters, and Group S (n=21), receiving intraoperative fluid management based on CVP (central venous pressure) parameters.

All patients in both groups will be encouraged to consume oral carbohydrate fluids (12.5% glucose solution) until two hours before surgery. Upon being brought to the operating table, routine electrocardiogram (ECG), peripheral oxygen saturation (SpO₂), end-tidal carbon dioxide (EtCO₂), and non-invasive blood pressure monitoring will be performed, and an 18G peripheral intravenous line will be placed. During surgery, all patients will receive a crystalloid infusion at 3 mL/kg/hour.

All patients will be intubated after intravenous induction with propofol (1.5-2 mg/kg), fentanyl (1-2 mcg/kg), and rocuronium (0.6 mg/kg). After induction, a 20G cannula will be placed in the radial artery of the upper extremity for monitoring. A 7 French triple-lumen central venous catheter will be placed in the right subclavian vein to manage potential complications. General anesthesia will be maintained with sevoflurane at approximately 1.0 (±20%) minimum alveolar concentration (MAC) with 40% FiO₂ (Fraction of Inspired Oxygen) at 1 L/min fresh gas flow. Both groups will be ventilated in volume-controlled mode with a tidal volume of 8 mL/kg. To calculate Crs in the supine position, a 10% inspiratory pause will be added to the ventilator settings to obtain plateau pressure. The surgery will be performed in the supine position, and the transducer will be positioned at the mid-axillary line in both groups. A urinary catheter will be inserted to monitor urine output. Additional doses of muscle relaxants and fentanyl will be administered as needed. NSAIDs, magnesium, and lidocaine will not be used to avoid affecting intraoperative hypotension or postoperative renal function. Intraoperative systolic arterial pressure will not be allowed to drop by more than 30% from baseline, and the mean arterial pressure will be maintained above 65 mmHg in normotensive patients and 80 mmHg in hypertensive patients. Hypotension will be defined as a drop of more than 20% from baseline mean arterial pressure.

According to institutional practice, 1 g/kg mannitol will be administered before the dura mater is opened. During dura mater opening, the surgical team will assess brain relaxation using a five-point scale (1=optimal conditions, 2=retraction not possible and dilated blood vessels, 3=tissue tension hindering intervention with obliterated sulci and dilated vessels, 4=worsening factors causing brain tissue extrusion, 5=worst conditions for surgery).

Patients with intraoperative hematocrit (Hct) <24% will receive erythrocyte suspension (ES). For patients with Hct >24%, transfusion will only occur with severe active bleeding. If Hct >24% and estimated blood loss is less than 10% of total blood volume, 1.5 times the amount of blood lost will be replaced with crystalloids. If Hct >24% and blood loss is estimated at 10-20% of total blood volume, 500 mL colloid will be administered. Blood loss will be estimated using the amount in the suction canister and the number of surgical sponges and gauzes used during surgery (a '4x4' gauze will be assumed to hold 10 mL, and a fully soaked laparotomy pad will be assumed to hold 150 mL of blood). In cases of severe volume deficit, colloids will be used to manage hypotensive periods until blood transfusion is administered. Diuresis will be targeted at 0.5 mL/kg/hour or higher in both groups.

In Group N, PPV values will be monitored continuously during the intraoperative period. If PPV >13%, patients will receive an additional 250 mL of crystalloid fluid over 10 minutes, followed by reevaluation. If PPV ≤13%, SBP <90 mmHg, MAP <65 mmHg, and HR <100 bpm, ephedrine will be administered. If more than 30 mg of ephedrine is required, dopamine infusion will be initiated. If PPV ≤13%, SBP <90 mmHg, MAP <65 mmHg, and HR >100 bpm, norepinephrine infusion will be used.

In Group S, CVP values will be monitored continuously. Patients will be disconnected from the ventilator for CVP measurement. If CVP <6 mmHg, patients will receive an additional 250 mL of crystalloid bolus over 10 minutes, followed by reevaluation. If CVP ≥6 mmHg, SBP <90 mmHg, MAP <65 mmHg, and HR <100 bpm, ephedrine will be administered. If more than 30 mg of ephedrine is required, dopamine infusion will be initiated. If CVP ≥6 mmHg, SBP <90 mmHg, MAP <65 mmHg, and HR >100 bpm, norepinephrine infusion will be used.

The demographic data of both groups (gender, age, BMI, ASA physical status classification score, comorbidities, baseline oxygen saturation (SpO₂), end-tidal carbon dioxide (EtCO₂), HR, MAP, CVP, PPV, creatinine, and serum lactate levels) and intraoperative data (surgery duration, fluid management protocol, postoperative creatinine and lactate levels, intraoperative hypotensive episodes, vasopressor requirements, volumes of crystalloids/colloids administered, number of bolus fluids given, volume of blood transfused, brain relaxation score, total intraoperative urine output) will be recorded.

Intraoperative SpO₂, EtCO₂, MAP, HR values, and hourly urine output of all patients will be recorded.

Fifteen minutes before the end of surgery, all patients will receive 100 mg tramadol and 1000 mg paracetamol in 150 mL normal saline as an IV infusion. At the end of surgery, 2-4 mg/kg sugammadex will be administered to reverse neuromuscular blockade. After extubation, patients will be transferred to the intensive care unit (ICU).

Postoperative creatinine and lactate levels will be measured and recorded at the 12th hour. The ICU length of stay will also be documented.

ELIGIBILITY:
Inclusion Criteria:

* ages of 18-65
* ASA (American Society of Anesthesiology) physical status classification score I-III
* who will undergo elective intracranial mass surgery under general anesthesia

Exclusion Criteria:

* Patients with renal failure
* mental retardation
* arrhythmia
* severe cardiopulmonary disease
* hemodynamic instability
* body mass index (BMI) >40 kg/m2
* respiratory system compliance (Crs) <30 mL/cmH2O
* use of lactate-producing drugs such as metformin
* lactate elevation at the beginning of the operation
* tumor causing diabetes insipitus
* patients who do not accept the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * ages of 18-65
  * ASA (American Society of Anesthesiology) physical status classification score I-III
  * who will undergo elective intracranial mass surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2024-04-03 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Fluid requirement (number of times needing bolus infusion-during surgery) | At 10-minutes intervals throughout the surgery
  Fluid requirement (number of times needing bolus infusion) One bolus infusion 250 mL amount
  Bolus fluid requirement will be assessed every 15 minutes throughout the operation.
  Assesment will make two method: CVP and PPV. Will be to compare the intraoperative fluid requirement between the two groups.
  1. CVP (Central Venous Pressure) group:
     In cases where CVP<6 mmHg during the intraoperative period, patients will be given an additional 250 ml bolus crystalloid infusion over a 10 minute period and LVB will be re-evaluated.
  2. PPV (Pulse Pressure Variation) group:
  In cases where the pulse pressure variations value is >13%, patients will be given an additional 250 ml of crystalloid fluid over a 10 minute period and pulse pressure variations will be reassessed.

SECONDARY OUTCOMES:
Duration of postoperative stay in the intensive care unit | in 2 weeks
  Evaluation of postoperative intensive care unit length of stay in days

OTHER OUTCOMES:
Intraoperative and postoperative creatinine value | Beginning of surgery, end of surgery and postoperative 24. hour creatinine value
  Creatinin value (Mg/dL)
  Intraoperative value (Beginning of surgery) Intraoperagive value (End of surgery) Postoperative 24. hour creatinine value
  All values will be compared between each other.
Intraoperative and postoperative serum lactate value | Beginning of the surgery, end of the surgery and postoperative 24. hour lactate value
  Serum lactate value (Mmol/L)
  Intraoperative lactate value (Beginning of the surgery) Intraoperagive lactate value (End of the surgery) Postoperative 24. hour lactate value
  All values will be compared between each other.
Brain relaxation scores | Within 5 minutes after surgical removal of the dura mater during surgery
  Brain relaxation scores will be evaluate middle of the surgery. Scores will be give from 1 to 5. During the opening of the dura mater, the surgical team will evaluate the brain relaxation with a five-point scale (Grade 1 - all factors are ideal, Grade 2 - retraction is not possible and blood vessels are dilated, Grade 3 - the tension of the brain tissue prevents the attempt, the sulci are erased together and the blood vessels are dilated, Grade 4 - these factors worsen and the brain tissue protrudes, Grade 5 - the worst conditions for surgery are present)
  Higher numbers mean worst outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Pamukkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I need to consider several factors when deciding whether or not to share Individual Participant Data (IPD). Privacy concerns are a primary issue, as ensuring the confidentiality of participants is critical. Additionally, the ethical constraints tied to the original consent process may limit sharing if explicit permissions were not obtained.

REFERENCES:
- [Background] Bristow A, Shalev D, Rice B, Lipton JM, Giesecke AH Jr. Low-dose synthetic narcotic infusions for cerebral relaxation during craniotomies. Anesth Analg. 1987 May;66(5):413-6. doi: 10.1213/00000539-198705000-00007. PMID 2953270
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Rail B, Hicks WH, Oduguwa E, Barrie U, Pernik MN, Montgomery E, Tao J, Kenfack YJ, Mofor P, Adeyemo E, Edukugho D, Caruso J, Bagley CA, El Ahmadieh TY, Aoun SG. Transfusion Guidelines in Brain Tumor Surgery: A Systematic Review and Critical Summary of Currently Available Evidence. World Neurosurg. 2022 Sep;165:172-179.e2. doi: 10.1016/j.wneu.2022.06.077. Epub 2022 Jun 23. PMID 35752421
- [Background] Gopal J, Srivastava S, Singh N, Haldar R, Verma R, Gupta D, Mishra P. Pulse Pressure Variance (PPV)-Guided Fluid Management in Adult Patients Undergoing Supratentorial Tumor Surgeries: A Randomized Controlled Trial. Asian J Neurosurg. 2023 Sep 22;18(3):508-515. doi: 10.1055/s-0043-1771364. eCollection 2023 Sep. PMID 38152505
- [Background] Vos JJ, Poterman M, Salm PP, Van Amsterdam K, Struys MM, Scheeren TW, Kalmar AF. Noninvasive pulse pressure variation and stroke volume variation to predict fluid responsiveness at multiple thresholds: a prospective observational study. Can J Anaesth. 2015 Nov;62(11):1153-60. doi: 10.1007/s12630-015-0464-2. Epub 2015 Sep 3. PMID 26335905
- [Background] Sundaram SC, Salins SR, Kumar AN, Korula G. Intra-Operative Fluid Management in Adult Neurosurgical Patients Undergoing Intracranial Tumour Surgery: Randomised Control Trial Comparing Pulse Pressure Variance (PPV) and Central Venous Pressure (CVP). J Clin Diagn Res. 2016 May;10(5):UC01-5. doi: 10.7860/JCDR/2016/18377.7850. Epub 2016 May 1. PMID 27437329
- [Background] Mayer J, Boldt J, Mengistu AM, Rohm KD, Suttner S. Goal-directed intraoperative therapy based on autocalibrated arterial pressure waveform analysis reduces hospital stay in high-risk surgical patients: a randomized, controlled trial. Crit Care. 2010;14(1):R18. doi: 10.1186/cc8875. Epub 2010 Feb 15. PMID 20156348
- [Background] Hofer CK, Muller SM, Furrer L, Klaghofer R, Genoni M, Zollinger A. Stroke volume and pulse pressure variation for prediction of fluid responsiveness in patients undergoing off-pump coronary artery bypass grafting. Chest. 2005 Aug;128(2):848-54. doi: 10.1378/chest.128.2.848. PMID 16100177
- [Background] Deflandre E, Bonhomme V, Hans P. Delta down compared with delta pulse pressure as an indicator of volaemia during intracranial surgery. Br J Anaesth. 2008 Feb;100(2):245-50. doi: 10.1093/bja/aem361. Epub 2007 Dec 14. PMID 18083787
- [Background] Montenij LJ, de Waal EE, Buhre WF. Arterial waveform analysis in anesthesia and critical care. Curr Opin Anaesthesiol. 2011 Dec;24(6):651-6. doi: 10.1097/ACO.0b013e32834cd2d9. PMID 22036950
- [Background] Teboul JL, Monnet X, Chemla D, Michard F. Arterial Pulse Pressure Variation with Mechanical Ventilation. Am J Respir Crit Care Med. 2019 Jan 1;199(1):22-31. doi: 10.1164/rccm.201801-0088CI. PMID 30138573
- [Background] Berkenstadt H, Margalit N, Hadani M, Friedman Z, Segal E, Villa Y, Perel A. Stroke volume variation as a predictor of fluid responsiveness in patients undergoing brain surgery. Anesth Analg. 2001 Apr;92(4):984-9. doi: 10.1097/00000539-200104000-00034. PMID 11273937
- [Background] Cannesson M, Le Manach Y, Hofer CK, Goarin JP, Lehot JJ, Vallet B, Tavernier B. Assessing the diagnostic accuracy of pulse pressure variations for the prediction of fluid responsiveness: a "gray zone" approach. Anesthesiology. 2011 Aug;115(2):231-41. doi: 10.1097/ALN.0b013e318225b80a. PMID 21705869
- [Background] Yang X, Du B. Does pulse pressure variation predict fluid responsiveness in critically ill patients? A systematic review and meta-analysis. Crit Care. 2014 Nov 27;18(6):650. doi: 10.1186/s13054-014-0650-6. PMID 25427970
- [Background] Voldby AW, Brandstrup B. Fluid therapy in the perioperative setting-a clinical review. J Intensive Care. 2016 Apr 16;4:27. doi: 10.1186/s40560-016-0154-3. eCollection 2016. PMID 27087980
- [Background] Marik PE, Cavallazzi R. Does the central venous pressure predict fluid responsiveness? An updated meta-analysis and a plea for some common sense. Crit Care Med. 2013 Jul;41(7):1774-81. doi: 10.1097/CCM.0b013e31828a25fd. PMID 23774337
- [Background] Gan TJ, Soppitt A, Maroof M, el-Moalem H, Robertson KM, Moretti E, Dwane P, Glass PS. Goal-directed intraoperative fluid administration reduces length of hospital stay after major surgery. Anesthesiology. 2002 Oct;97(4):820-6. doi: 10.1097/00000542-200210000-00012. PMID 12357146
- [Background] Bellamy MC. Wet, dry or something else? Br J Anaesth. 2006 Dec;97(6):755-7. doi: 10.1093/bja/ael290. No abstract available. PMID 17098724
- [Background] Miller TE, Myles PS. Perioperative Fluid Therapy for Major Surgery. Anesthesiology. 2019 May;130(5):825-832. doi: 10.1097/ALN.0000000000002603. No abstract available. PMID 30789364